CLINICAL TRIAL: NCT05385081
Title: PREcision Medicine in Cancer in Odense, Denmark (PRECODE) Feasibility of Genomic Profiling and Frequency of Genomic Matched Treatment in Solid Tumors With no Treatment Options
Brief Title: PREcision Medicine in Cancer in Odense, Denmark
Acronym: PRECODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karin Holmskov Hansen, MD, Principal Investigator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRECODE_S-20180147G
Record Dates: First submitted 2022-01-07; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Genetic Profile

STUDY DESIGN:
Intervention Model Description: prospective, single-center cohorte study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- genomic profiling (Other): After informed consent a PET/CT scan is performed to determine disease spread and the best location for core needle biopsi. Genomic profiling is performed using Next Generation Sequencing, NGS, genpanel analysis by Oncomine Comprehensive vs 3 The result of NGS is discussed at weekly local and national tumor board meeting to decide a possible targeted treatment offer based on genomic profiling or a possibly treatment offer in a clinical trial.
  Timelines in the course of investigation will be calculated using date of informed consent, PET/CT scan, biopsy, tumor board and date of start of next treatment, progression and death.
  If the genomic profiling results in a targeted treatment offer the Growth Modulation Index is calculated from progressions-free survival on recent and current treatment. Treatment given without an actionable target is likewise evaluated for efficacy.
  Interventions: Other: genomic profiling

INTERVENTIONS:
Other: genomic profiling — next generation sequencing

SUMMARY:
The traditional approach to cancer treatment has changes from using drugs approved for the specific cancer diagnosis to a tumor agnostic approach when treating solid tumors. How often will tumor biopsy and genomic profiling in patients with advanced solid tumors with no further evidence based treatment options result in biomarker-driven targeted treatment ? Feasibility of the investigation of patients and median turnaround time from biopsy to available genomic profile is evaluated.

DETAILED DESCRIPTION:
Genomic profiling in patients with advanced solid tumors and no further evidence based treatment options is a newer approach. The frequency of genomic alterations varies between individual tumor types and the actionability of somatic variants are different but evolves in line with the development of new targeted drugs. In accordance with expected short survival short assessment time is important to minimize the risk of patient detoriation during the investigation. A fresh biopsy from lesions in progression is preferred for analysis. To minimize the duration of the genomic profiling a genpanel analysis covering the most frequent oncogene targets is preferred.

The primary objective is to evaluate the feasibility of the investigational procedures. The secondary objective is to investigate how often genomic changes in tumor tissue gives rise to a targeted treatment offer and to evaluate the clinical benefit using the Growth Modulation Index.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Diagnosis of advanced solid tumors
* Evidence based treatment options are exhausted
* Performance Status 0-2
* Adequate organ function
* Life expectancy of at least 3 months

Exclusion Criteria:

• inclusions criteria not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Turn around time genomic profiling | through study completion, an average of 2 year
  Time from date of biopsi to date of available genomic profile discussed at tumor board meeting

SECONDARY OUTCOMES:
Frequenc of matched treatment offer | through study completion, an average of 2 year
  Number of patients offered a treatment based on the genomic profile

CONTACTS AND LOCATIONS:
Overall Officials: Karin H Hansen, Principal Investigator — Departement of Oncology Odense University Hospital
Locations (1):
- Odense Universitets Hospital dept of oncology, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen KH, Lyng MB, Kodahl AR, Asmussen JT, Arshad A, Petersen H, Krogh L, Ehmsen S, Kristensen TK, Ditzel HJ. Genomic profiling and expanded use of targeted anticancer drugs in solid cancers with exhausted evidence-based treatment options (PRECODE): study protocol of a prospective, non-randomized, cohort study. BMC Med Genomics. 2024 Nov 21;17(1):274. doi: 10.1186/s12920-024-02033-z. PMID 39574115